CLINICAL TRIAL: NCT03836365
Title: Patient Preparedness for Pelvic Organ Prolapse Surgery: A Randomized Controlled Trial of Preoperative Counseling
Brief Title: Patient Preparedness for Pelvic Organ Prolapse Surgery
Acronym: PREOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, Jessica Sassani, Fellow, Division of Female Pelvic Medicine & Reconstructive Surgery, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY19010073
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Pelvic Organ Prolapse; Patient Preparedness
Keywords: Pelvic organ prolapse; Patient preparedness; Randomized controlled trial
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Working Conditions; CD56 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative counseling office visit (Active Comparator): Participants will present for an in-person preoperative counseling office visit (preoperative counseling session). This will occur within a few weeks of surgery. Preoperative counseling topics are standardized and will be identical with each arm.
  Interventions: Other: Preoperative counseling office visit
- Preoperative counseling phone call (Active Comparator): Participants will receive a preoperative counseling phone call (preoperative counseling session). This will occur within a few weeks of surgery. Preoperative counseling topics are standardized and will be identical with each arm.
  Interventions: Other: Preoperative counseling phone call

INTERVENTIONS:
Other: Preoperative counseling office visit — All patients undergo a preoperative counseling session prior to surgery. Participants in this arm will have an in person preoperative counseling office visit.
  Other Names: Office
  Arms: Preoperative counseling office visit
Other: Preoperative counseling phone call — All patients undergo a preoperative counseling session prior to surgery. Participants in this arm will have a preoperative counseling phone call.
  Other Names: Call
  Arms: Preoperative counseling phone call

SUMMARY:
Patient preparedness has been associated with increased patient satisfaction, decreased postoperative pain and decreased postoperative narcotic use; however, little is known regarding the optimal way to prepare patients prior to pelvic reconstructive surgery. The primary aim of this study is to determine if a preoperative counseling in person visit has similar rates of patient preparedness as a preoperative counseling phone call for women undergoing same-day pelvic organ prolapse surgery. Secondary aims evaluate patient satisfaction, postoperative pain scores and postoperative narcotic usage. Women who plan to undergo pelvic organ prolapse surgery will be randomized to a preoperative in person counseling visit or a preoperative counseling phone call. Participants will complete questionnaires to assess their preparedness, satisfaction and postoperative pain. The goal of this study is to gather information that will allow clinicians to improve patient surgical preparedness and satisfaction.

DETAILED DESCRIPTION:
This will be a randomized controlled trial to assess patient preparedness following a preoperative counseling in person visit when compared to a preoperative counseling phone call.

Recruitment & Enrollment: Participants will be recruited and enrolled from the urogynecology office during their surgical planning visit. The study will be introduced at this visit and participants will have the opportunity to bring the consent home to review and consider their participation prior to signing.

Randomization: Participants will be block randomized in a 1:1 ratio in block size of 2. Randomization will be done by REDCap. The participant will not be blinded given the nature of the intervention. Additionally, the attending surgeon, fellow and office staff (advanced practice providers, research staff, medical assistants) will be aware of the randomization group as they will be participating in the preoperative intervention or perioperative clinical care.

Intervention: Both the preoperative counseling visit and preoperative phone call will contain the same components of discussion and counseling which include surgical details, risks and benefits, preoperative and postoperative instructions and expectations. The visit will take place in the urogynecology office and the visits and phone calls will be done by either a fellow or advanced practice provider, all of whom have extensive experience with the standardized preoperative visit.

Follow up: A postoperative phone call will be completed either POD#1 or POD#2 to remind the participant to complete their daily pain diary. Each participant will follow up for their standard postoperative visit approximately 4-6 weeks postoperative. All patients routinely receive a call on POD#1 from our nurses to assess how they are doing postoperatively. This phone call will continue unchanged for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Women planning to undergo same-day surgery to correct pelvic organ prolapse by the University of Pittsburgh Division of Urogynecology. Women remain eligible if they are admitted for observation following their surgery.

Exclusion Criteria:

* Non-English speaking patients
* A preoperative exam requirement that would necessitate an in person office visit (i.e. need for pessary removal, self-catheterization teaching)
* Plan for concomitant surgical management with gynecology oncology or colorectal surgery
* Residence in a nursing home

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Patient preparedness | At postoperative visit (about 4-6 weeks after surgery)
  The percent of patients reporting preparedness on Preoperative Preparedness Questionnaire. Participants who answer "strongly agree" or "agree" to the statement "Overall, I felt prepared for my surgery" will be considered prepared. This instrument is a 9-item questionnaire and scored on a 5-point Likert scale with answers ranging from "5=strongly disagree" to "1=strongly agree" with "3=neutral." Therefore, scores of "1=strongly agree" or "2=agree" will be considered a positive answer for preparedness. It was adopted from a study by Kenton et al in 2007.

SECONDARY OUTCOMES:
Patient satisfaction: Decision Scale-Pelvic Floor Disorders questionnaire | At postoperative visit (about 4-6 weeks after surgery)
  The percent of patients reporting satisfaction on the Satisfaction with Decision Scale-Pelvic Floor Disorders questionnaire. This is a validated, 5-item questionnaire with answers on a 5-point likert scale with "1=strongly agree," "3=neutral" and "5=strongly disagree." Answers of "1=strongly agree" or "2=agree" to the statement "I am satisfied with my decision" will be considered satisfied.
Postoperative pain scores | Postoperative days #1-7
  Postoperative pain scores on postoperative days #1-7 on a scale of 0-10. Participants will complete a daily pain diary which will assess their pain score with 0=no pain and 10=worst pain imaginable.
Postoperative narcotic use | Postoperative days #1-7
  Postoperative narcotics used which will be assessed by the daily pain diary (question: "How many narcotic pills did you use today?" with the answer being the number of pills used that day).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Sassani, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens' Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers

REFERENCES:
- [Background] Holmes-Rovner M, Kroll J, Schmitt N, Rovner DR, Breer ML, Rothert ML, Padonu G, Talarczyk G. Patient satisfaction with health care decisions: the satisfaction with decision scale. Med Decis Making. 1996 Jan-Mar;16(1):58-64. doi: 10.1177/0272989X9601600114. PMID 8717600
- [Background] Sung VW, Kauffman N, Raker CA, Myers DL, Clark MA. Validation of decision-making outcomes for female pelvic floor disorders. Am J Obstet Gynecol. 2008 May;198(5):575.e1-6. doi: 10.1016/j.ajog.2007.12.035. Epub 2008 Mar 7. PMID 18313632
- [Result] Kenton K, Pham T, Mueller E, Brubaker L. Patient preparedness: an important predictor of surgical outcome. Am J Obstet Gynecol. 2007 Dec;197(6):654.e1-6. doi: 10.1016/j.ajog.2007.08.059. PMID 18060968